CLINICAL TRIAL: NCT05251974
Title: The Effect of Medication Compliance, Verified With Medication Level Testing, on Unplanned Hospital Readmission or Urgent Outpatient Visit in Patients With Acute Decompensated Heart Failure
Brief Title: Assay to Measure Beta Blocker Adherence
Status: Terminated | Type: Observational
Why Stopped: Quest Diagnostics terminated study early - did not want to continue to support single-site study
Sponsor: Summa Health System (Other)
Collaborators: Quest Diagnostics-Nichols Insitute (Industry)
Responsible Party: Sponsor
Other Study IDs: 21145
Record Dates: First submitted 2022-02-11; First posted 2022-02-23 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Congestive Heart Failure; Medication Adherence
MeSH Terms: conditions — Heart Failure; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Compliant with beta blocker therapy: Patients observed to be compliant with beta blocker therapy by blood assay
  Interventions: Diagnostic Test: Quest beta blocker assay
- Non-compliant with beta blocker therapy: Patients observed to be non-compliant with beta blocker therapy by blood assay
  Interventions: Diagnostic Test: Quest beta blocker assay

INTERVENTIONS:
Diagnostic Test: Quest beta blocker assay — Blood assay to detect presence of beta blocker medications

SUMMARY:
This study will assess the feasibility and efficacy of using serum assay developed by Quest Diagnostics to detect the presence of beta blockers, specifically carvedilol and metoprolol succinate, in patients with heart failure.

DETAILED DESCRIPTION:
Patients admitted to the Summa Akron City campus with a primary diagnosis of heart failure will be invited to participate 1 to 2 days prior to expected discharge. A research nurse with the Summa CRC will enroll patients, obtain informed consent, and perform all study-related blood sample collection. We will collect blood from each enrolled patient up to three times. The first blood sample collection will be obtained just prior to discharge. A second and third blood sample will be collected at the patient's routine 7-day and 30-day post-hospital follow up appointment, respectively. Each blood draw will collect 13mL of blood from each patient, for a total of up to 39mL of blood for the entire study. If the patient is readmitted for heart failure prior to the 7- or 30-day follow up appointment, the subsequent blood draws will be cancelled.

Our enrollment target is 100 patients. Patients admitted to the Summa Akron City campus with a primary diagnosis of heart failure will be invited to participate 1 to 2 days prior to expected discharge. A research nurse with the Summa CRC will enroll patients, obtain informed consent, and perform all study-related blood sample collection. We will collect blood from each enrolled patient up to three times. The first blood sample collection will be obtained just prior to discharge. A second and third blood sample will be collected at the patient's routine 7-day and 30-day post-hospital follow up appointment, respectively. Each blood draw will collect 13mL of blood from each patient, for a total of up to 39mL of blood for the entire study. If the patient is readmitted for heart failure prior to the 7- or 30-day follow up appointment, the subsequent blood draws will be cancelled.

Additionally, study personnel will asses medication adherence at the 7- and 30-day follow up appointments by asking the patient 1) if they took their most recent scheduled dose of their beta blocker, and 2) how often do they miss their scheduled beta blocker dose. Study personnel will also verify medication list and record other cardiology medications used at the 7- and 30-day follow ups. Blood samples will be labeled with the study code and patient DOB, and sent to Quest Diagnostics via courier for analysis. Date/time for each blood sample will be recorded. This information will be recorded on the Quest Visit Worksheet which will be stored in the subjects study binder. For each blood sample, Quest will quantify the amount of beta blocker present, as well as creatinine, and NT-proBNP level present. The patient's providers will be blinded to the assay results until after the 30-day study period has elapsed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-89
* Admitted for primary diagnosis of heart failure with reduced ejection fraction
* Prescribed carvedilol or metoprolol succinate for beta blocker therapy
* Will be following up at 95 Arch St. Clinic

Exclusion Criteria:

* Under age 18/over age 89
* Patients that plan to follow up somewhere other than the 95 Arch St. Clinic
* Patients with prior heart transplant or a left ventricular assist device
* Patient is unable to provide consent.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized with a primary diagnosis of heart failure with reduced ejection fraction at Summa Health - Akron Campus.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Readmission/urgent outpatient visit | 30 days
  Requiring readmission or an urgent outpatient visit for heart failure

SECONDARY OUTCOMES:
Mortality | 30 days
  All-cause mortality during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Varian, MD, Principal Investigator — Summa Health System
Locations (1):
- Summa Health System, Akron, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
N/A - no plan to make IPD available.